CLINICAL TRIAL: NCT00541424
Title: Feasibility of Combined CT Colonography and PET Imaging for Detection of Colonic Involvement by Mantle Cell Lymphoma
Brief Title: Combined CT Colonography and PET Imaging in Mantle Cell Lymphoma
Status: Withdrawn | Type: Observational
Why Stopped: No study recruitment due to time constraints and lack of support.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1112
Record Dates: First submitted 2007-10-08; First posted 2007-10-10 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Mantle Cell Lymphoma; Lymphoma
Keywords: Mantle Cell Lymphoma; Lymphoma; CT Colonography; PET Scan; PET/CT Scan; Gas Insufflation
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT Scanning: Patients that have newly diagnosed mantle cell lymphoma will first undergo CT colonography (CT or CTC) and PET followed by conventional colonoscopy.
  Interventions: Procedure: PET/CT Scanning

INTERVENTIONS:
Procedure: PET/CT Scanning — Full-body PET/CT procedure will be performed. Gas will be pumped into the colon before the scan so the colon will be opened up (inflated) and the study doctor will be able to more easily look for any lesions. This procedure is called gas insufflation.

SUMMARY:
The goal of this clinical research study is to learn if positron emission tomography (PET)/computed tomography (CT) scanning can be used to detect mantle cell lymphoma in the colon. Researchers want to learn if PET/CT scanning can produce good-quality images and/or find the exact locations of lymphoma in the body.

Primary Objective is to determine if combined CT colonography and full body PET scan is technically feasible and can produce diagnostic scans as well as accurate anatomic coordination for detection of mantle cell lymphoma involvement of the colon.

DETAILED DESCRIPTION:
Colonoscopy Testing:

A colonoscopy is a routine test where the doctor looks at the inner lining of the colon using a long, flexible, lighted tube that is inserted through the anus. This is the standard procedure for detecting mantle cell lymphoma in the colon.

PET/CT Scanning:

Because PET/CT scanning is less invasive than colonoscopy, researchers want to learn more about whether PET/CT scanning may be able to be used for detecting mantle cell lymphoma in the colon.

PET/CT scanning is also considered a routine test for checking the status of mantle cell lymphoma. The scan is called "full body" because the neck, chest, abdomen (stomach area), and pelvis are included.

In this study, participants will have a full-body PET/CT procedure performed like they normally would, but the difference will be that gas will be pumped into the colon before the scan. This is so the colon will be opened up (inflated) so the study doctor will be able to more easily look for any lesions. The procedure is called gas insufflation. (In standard PET/CT scanning of the colon, gas insufflation is not used.)

Study Participation:

If you agree to take part in this study, you will begin the PET/CT procedure, as usual. This means a special substance called fluorodeoxyglucose will be injected by vein, in order to make the tumor more visible in the scanned image.

About an hour later, the study doctor will prepare your colon for the PET/CT scan by performing gas insufflation. To do so, a soft plastic tube will be inserted through your anus. Carbon dioxide gas will be automatically pumped into your colon until the gas is at the correct pressure.

If the study doctor decides it is necessary (for example, if cramping occurs), you will receive a glucagon injection under the skin in order to relax the colon. Glucagon is a medication that helps to relax the colon and decrease cramping. If continued cramping occurs, the gas will be turned off which results in immediate relief. This is considered routine for the CT part of the PET/CT. Administering the gas for the CT is similar to the sensation that will be felt during the colonoscopy when the colon is also insufflated.

After the gas insufflation, the routine PET/CT scan will be performed to check the status of the disease. You will lie on your stomach for the first part of the PET/CT scan and on your back for the second part.

After the PET/CT scan, the routine colonoscopy will be performed. You will need to sign a separate consent form for the colonoscopy, and the procedure will be explained to you in detail.

Length of Study:

Your participation in this study will be over after the PET/CT scan. Researchers will compare the results of the PET/CT scan to the results of the colonoscopy.

This is an investigational study. Gas insufflation and glucagon are FDA approved for use with CT colonography (colonoscopy that uses CT scanning), which is typically used to screen for colon cancer. PET/CT scanning is FDA approved for use in checking the status of mantle cell lymphoma. Using PET/CT scanning to detect mantle cell lymphoma in the colon, however, is investigational. For this purpose, at this time PET/CT scanning is being used in research only.

Up to 43 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have newly diagnosed mantle cell lymphoma who are already scheduled for standard PET/CT and colonoscopy as part of their staging.
* Adults (>18 years of age)

Exclusion Criteria:

* Known diabetes
* Known complete colonic obstruction
* Known small bowel obstruction
* Known anorectal stenosis or acute inflammatory disease or rectal prolapse.
* Active colitis or diverticulitis
* Known radiation in the last 2 weeks
* Known endoscopic hot forceps biopsy in the last 2 weeks
* Known rectal incontinence
* Tachypnea or respiratory distress
* Known end or loop colostomy or ileostomy
* Contraindications to colonoscopy, including bleeding diathesis; contraindications to sedation because of allergy or respiratory compromise.
* Patients who are pregnant
* Diarrhea within the past week
* Currently participating in chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have newly diagnosed mantle cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of Participants with PET/CT Scan Detection of Mantle Cell Lymphoma | 1 Day, Participation completed day of CT colonography and full body PET scan

SECONDARY OUTCOMES:
Number of PET/CT Scanning Images Locating Exact Lymphoma Locations | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Revathy B. Iyer, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org